CLINICAL TRIAL: NCT02892201
Title: A Phase II Study of Pembrolizumab for Patients With Head and Neck Squamous Cell Carcinoma With Residual Disease Following Definitive Chemoradiation
Brief Title: Pembrolizumab in HNSCC With Residual Disease After Radiation
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Low enrollment
Sponsor: Yale University (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2000028047; 1602017275 (Other: Original Yale IRB ID)
Record Dates: First submitted 2016-08-19; First posted 2016-09-08 (Estimated); Results first posted 2023-11-18 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-07

CONDITIONS: Head and Neck Squamous Cell Carcinoma
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- All subjects (Experimental): for patients with squamous cell carcinoma of the head and neck who have residual disease following definitive therapy with radiation
  Pembrolizumab will be given at a constant dose of 200 mg every three weeks, for four cycles. Patients with resectable disease can then go on to surgery, and patients with unresectable disease can continue on pembrolizumab until progression or for up to 1 year.
  Interventions: Drug: Pembrolizumab

INTERVENTIONS:
Drug: Pembrolizumab — a constant dose of 200 mg every three weeks, for four cycles.
  Other Names: Keytruda; MK-3475

SUMMARY:
This is a phase II study for patients with squamous cell carcinoma of the head and neck who have residual disease following definitive therapy with radiation (with or without systemic therapy). Patients must be diagnosed with residual disease within 24 weeks of completion of radiation therapy. Residual disease must be biopsy proven before the patient can consent to the trial, and can be either from lymph nodes in the neck, or from the primary tumor site. Prior to beginning study therapy patients are evaluated by an ENT to determine if they have disease amenable to surgical resection. Both resectable and unresectable patients will be eligible for participation in the study.

DETAILED DESCRIPTION:
The primary objective is to determine the overall response to pembrolizumab for patients with residual disease following radiation with or without systemic therapy for squamous cell carcinoma of the head and neck.

Hypothesis: The use of pembrolizumab in patients with residual disease following radiation with or without systemic therapy will lead to an enhanced overall response rate due to treatment-related priming of the immune response.

When initially registered, the study used a follow up assessment of 12 weeks. However, the actual study aims for the primary and secondary outcomes were updated to 168 weeks. The primary completion date was also updated to reflect the primary outcome timeline.

Following results entry and QC review, the Overall Response Rate at 168 weeks secondary outcome, defined as a composite of 2 measures, was removed as it was reported in separate outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Be willing and able to provide written informed consent/assent for the trial.
2. Be => 18 years of age on day of signing informed consent.
3. Biopsy proven residual disease.
4. Be willing to provide tissue from a newly obtained core biopsy of a tumor lesion. Newly-obtained is defined as a specimen obtained up to 6 weeks (42 days) prior to initiation of treatment on Day 1 and following completion of RT/CRT.
5. Have a performance status of 0 or 1 or 2 on the ECOG Performance Scale.
6. Demonstrate adequate organ function. Labs value need to be assessed within 14 days of study treatment.
7. Female subject of childbearing potential should have a negative urine or serum pregnancy within 72 hours prior to receiving the first dose of study medication. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
8. Female subjects of childbearing potential should be willing to use 2 methods of birth control or be surgically sterile, or abstain from heterosexual activity for the course of the study through 120 days after the last dose of study medication (Reference Section 5.7.2). Subjects of childbearing potential are those who have not been surgically sterilized or have not been free from menses for > 1 year.
9. Male subjects should agree to use an adequate method of contraception starting with the first dose of study therapy through 120 days after the last dose of study therapy.
10. Patients must have a history of Stage I-IVB SCC of the head and neck arising from the oral cavity, oropharynx, nasopharynx, larynx, or hypopharynx and must have been treated with definitive intent radiation (with or without systemic therapy)
11. Patients must be at least 6 weeks (42 days) and no more than 24 weeks (168 days) from completion of radiation with or without systemic therapy at the time of biopsy confirming residual disease. Patients must receive the first dose of study medication no more than 28 weeks following completion of radiation.
12. Patients must have pathological evidence of persistent lymph node disease or persistent disease at the primary tumor site with viable tumor cells confirmed by a biopsy within 24 weeks of study treatment and no evidence of metastatic disease following primary radiation with or without systemic therapy confirmed by a CT scan within 4 weeks of study treatment. If a biopsy confirming residual disease has not been performed, this can be performed after obtaining consent during the screening procedures.
13. Persistent lymph node disease with viable tumor cells will be determined by the histological determination of tumor viability.
14. All persistent disease must have received at least 66 Gy in 1.8-2Gy fractions of radiotherapy to the area of residual disease (or a biologically equivalent dose given by the linear quadratic equation: biologically equivalent dose (BED) = nd (1 + d/( α/β), where n is the number of fractions, d dose per fraction and the α/β ratio for tumor is 10. Previous radiation records will be obtained to confirm adequate dosing.

Exclusion Criteria:

1. Is currently participating and receiving study therapy or has participated in a study of an investigational agent and received study therapy or used an investigational device within 4 weeks of the first dose of treatment.
2. Has a diagnosis of immunodeficiency or is receiving supraphysiologic doses of systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment. A physiologic dose of steroids is defined as up to 10mg of prednisone daily (or its equivalent).
3. Has a known history of active TB (Bacillus Tuberculosis)
4. Hypersensitivity to pembrolizumab or any of its excipients.
5. Has had a prior anti-cancer monoclonal antibody (mAb) within 4 weeks prior to study Day 1 or who has not recovered (i.e., ≤ Grade 1 or at baseline) from acute, non-hematological adverse events due to agents administered more than 4 weeks earlier, unless otherwise approved by the Principal Investigator.

   * Note: Subjects with ≤ Grade 2 neuropathy, any grade dysphagia, ≤ Grade 2 pain, ≤ Grade 2 weight loss, any grade hyperpigmentation of skin, any grade fatigue, any grade xerostomia, and any grade dysgeusia, are an exception to this criterion and may qualify for the study. Also please note that the presence of a feeding tube to aid with nutrition does not disqualify patients from study.
   * Note: If subject received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy.
6. Has had prior chemotherapy, targeted small molecule therapy, or radiation therapy within 2 weeks prior to the first protocol treatment or who has not recovered (i.e., ≤ Grade 1 or at baseline) from acute, non-hematological adverse events due to a previously administered agent, unless otherwise approved by the Principal Investigator.

   * Note: Subjects with ≤ Grade 2 neuropathy, any grade dysphagia, ≤ Grade 2 pain, ≤ Grade 2 weight loss, any grade hyperpigmentation of skin, any grade fatigue, any grade xerostomia, and any grade dysgeusia, are an exception to this criterion and may qualify for the study. Also please note that the presence of a feeding tube to aid with nutrition does not disqualify patients from study.
   * Note: If subject received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy.
7. Has a known additional malignancy that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin or squamous cell carcinoma of the skin that has undergone potentially curative therapy or in situ cervical cancer.
8. Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis. Subjects with previously treated brain metastases may participate provided they are stable (without evidence of progression by imaging for at least four weeks prior to the first dose of trial treatment and any neurologic symptoms have returned to baseline), have no evidence of new or enlarging brain metastases, and are not using steroids for at least 7 days prior to trial treatment. This exception does not include carcinomatous meningitis which is excluded regardless of clinical stability.
9. Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (eg., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
10. Has known history of non-infectious pneumonitis that required steroids, or current pneumonitis.
11. Has an active infection requiring systemic therapy.
12. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
13. Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
14. Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 120 days after the last dose of trial treatment.
15. Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti-PD-L2 agent.
16. Has a known history of Human Immunodeficiency Virus (HIV) (HIV 1/2 antibodies).
17. Has known active Hepatitis B (e.g., HBsAg reactive) or Hepatitis C (e.g., HCV RNA [qualitative] is detected).
18. Has received a live vaccine within 30 days of the first protocol treatment. Note: Seasonal influenza vaccines for injection are generally inactivated flu vaccines and are allowed; however intranasal influenza vaccines (e.g., Flu-Mist®) are live attenuated vaccines, and are not allowed.
19. Any patient receiving adjuvant systemic therapy following the completion of radiation therapy is ineligible.
20. Any patient with evidence of distant metastatic disease on a CT within 4 weeks of treatment is ineligible.
21. Evidence of interstitial lung disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2016-09-08 (Actual); Primary Completion 2020-02 (Actual); Study Completion 2020-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Burtness, MD, Principal Investigator — Yale University
Locations (2):
- United States (2):
  - Yale Cancer Center, New Haven, Connecticut
  - University of Texas Southwestern Medical Center (UTSW), Dallas, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study was activated for enrollment on 9/08/2016 and was closed for low enrollment on 03/31/2020.
  Enrollment done in a medical Clinic.
Groups:
- All Subjects: For patients with squamous cell carcinoma of the head and neck who have residual disease following definitive therapy with radiation
  Pembrolizumab will be given at a constant dose of 200 mg every three weeks, for four cycles. Patients with resectable disease can then go on to surgery, and patients with unresectable disease can continue on pembrolizumab until progression or for up to 1 year.
  Pembrolizumab: a constant dose of 200 mg every three weeks, for four cycles.
Period: Overall Study
Arm/Group | All Subjects
Started | 9 (For purpose of the primary endpoint of the study, the overall response will be measured during the post pembrolizumab, in comparison to the most immediate pre-pembrolizumab imaging.)
Completed | 9
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | All Subjects
Number analyzed (Participants) | 9
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 3
  >=65 years | 6
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 8
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 6
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 9

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate
Description: To determine the overall response rate based on RECIST 1.1 to pembrolizumab for patients with residual disease following radiation with or without systemic therapy for squamous cell carcinoma of the head and neck. For lesions considered too small for measurement by RECIST 1.1 a modified response criteria will be used. RECIST categories used for the target lesion are complete response (CR), partial response (PR), stable disease (NR/SD), and progressive disease (PD). Upon entry of results, the time frame was corrected to 12 weeks (see attached protocol).
Time Frame: 12 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | All Subjects
Number analyzed (Participants) | 9
Participants
  complete response (CR) | 1
  partial response (PR) | 1
  stable disease (SD) | 0
  progressive disease (PD) | 7

2. Secondary Outcome: Change in PD-L1 Expression
Description: To determine changes in PD-L1 expression following irradiation, the Modified Proportion Score or MPS was used. MPS is a scale of 0-100 and it represents the overall % positive cells expressing PD-L1 where the greater the score, the more likely there will be a response to treatment. This outcome was updated/corrected at the time of results entry.
Time Frame: Up to 4 weeks
Population: 6 total participants had evaluable data at baseline, 2 had evaluable data at the 4 week follow up and 1 person withdrew consent at follow up.
Measure: Median (Full Range); unit: score on a scale
Arm/Group | All Subjects
Number analyzed (Participants) | 6
score on a scale
  Baseline | 25.5 [0 to 90]
  Week 4: number analyzed (Participants) | 2
  Week 4 | 7.5 [0 to 15]
  Baseline to Week 4 Change on Matched Cases: number analyzed (Participants) | 2
  Baseline to Week 4 Change on Matched Cases | 17.5 [0 to 35]

3. Secondary Outcome: Median Progression Free Survival
Description: To evaluate median progression free survival in days. Upon entry of results, the time frame was corrected to the full amount of time that participants were followed up with.
Time Frame: Up to 168 weeks
Measure: Median (Full Range); unit: days
Arm/Group | All Subjects
Number analyzed (Participants) | 9
days | 74 [14 to 1902]

4. Secondary Outcome: Overall Survival
Description: To evaluate overall survival. Overall survival is presented as a count of those deceased and living at the end of the follow up period.
Time Frame: 168 weeks
Population: 1 person withdrew consent for long term follow up.
Measure: Count of Participants; unit: Participants
Arm/Group | All Subjects
Number analyzed (Participants) | 8
Participants
  Confirmed Deceased | 5
  Confirmed Living | 3

5. Secondary Outcome: Median Overall Survival
Description: To evaluate overall survival, the median overall survival time is presented in days through the study and follow up periods.This outcome was reported at the time of results entry to compliment the count of participants in the Overall Survival outcome.
Time Frame: Up to 168 weeks
Population: 1 person withdrew consent for long term follow up.
Measure: Median (Full Range); unit: days
Arm/Group | All Subjects
Number analyzed (Participants) | 8
days | 505 [243 to 1905]

6. Other Pre Specified Outcome: Count of Participants With Immune Related Adverse Events
Description: To determine the number of participants receiving immunotherapy following radiation with or without systemic therapy. This outcome was updated/corrected at the time of results entry.
Time Frame: 12 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | All Subjects
Number analyzed (Participants) | 9
Participants
  Experienced immune related adverse event | 4
  Did not experience an immune related adverse event | 5

7. Other Pre Specified Outcome: Count of Those With Distant Metastases
Description: Presented are a count of those that experienced distant metastases during the study period and follow up period. This outcome was updated/corrected when results were entered.
Time Frame: 168 Weeks
Population: 1 participant withdrew consent for follow up.
Measure: Count of Participants; unit: Participants
Arm/Group | All Subjects
Number analyzed (Participants) | 8
Participants
  Distant Metastases: YES | 1
  Distant Metastases: NO | 7

8. Other Pre Specified Outcome: Overall Response Rate
Description: To determine the overall response rate based on RECIST 1.1 to pembrolizumab for patients with residual disease following radiation with or without systemic therapy for squamous cell carcinoma of the head and neck. For lesions considered too small for measurement by RECIST 1.1 a modified response criteria will be used. RECIST categories used for the target lesion are complete response (CR), partial response (PR), stable disease (NR/SD), and progressive disease (PD). This outcome was originally incorrectly listed as a secondary outcome.
Time Frame: 168 weeks
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Up to 168 weeks
Arm/Group | All Subjects
All-Cause Mortality (participants affected / at risk) | 5/9
Serious Adverse Events (participants affected / at risk) | 6/9
Other Adverse Events (participants affected / at risk) | 8/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Subjects (N=9)
Cardiac disorders - Other, specify (Cardiac disorders) | 1 (1)
Myocardial infarction (Cardiac disorders) | 1 (1)
Oral hemorrhage (Gastrointestinal disorders) | 1 (1)
Upper respiratory infection (Infections and infestations) | 1 (1)
Hematuria (Renal and urinary disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Laryngeal edema (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pharyngeal hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypertension (Vascular disorders) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 1 (1)
Hypotension (General disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Subjects (N=9)
Anemia (Blood and lymphatic system disorders) | 1 (1)
Blood and lymphatic system disorders - Other, specify (Blood and lymphatic system disorders) | 1 (2)
Hemolytic uremic syndrome (Blood and lymphatic system disorders) | 1 (1)
Thrombotic thrombocytopenic purpura (Blood and lymphatic system disorders) | 1 (1)
Cardiac disorders - Other, specify (Cardiac disorders) | 1 (1)
Ear pain (Ear and labyrinth disorders) | 1 (1)
Hypothyroidism (Endocrine disorders) | 2 (2)
Constipation (Gastrointestinal disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 2 (2)
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (2)
Periodontal disease (Gastrointestinal disorders) | 1 (1)
Fatigue (General disorders) | 3 (4)
General disorders and administration site conditions - Other, specify (General disorders) | 4 (16)
Localized edema (General disorders) | 1 (1)
Neck edema (General disorders) | 1 (1)
Infections and infestations - Other, specify (Infections and infestations) | 1 (1)
Bruising (Injury, poisoning and procedural complications) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1)
Alkaline phosphatase increased (Investigations) | 2 (4)
Aspartate aminotransferase increased (Investigations) | 1 (1)
Creatinine increased (Investigations) | 1 (1)
Lymphocyte count decreased (Investigations) | 2 (3)
Platelet count decreased (Investigations) | 1 (1)
Weight loss (Investigations) | 3 (5)
White blood cell decreased (Investigations) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 2 (4)
Hypoglycemia (Metabolism and nutrition disorders) | 1 (1)
Hypomagnesemia (Metabolism and nutrition disorders) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Nervous system disorders - Other, specify (Nervous system disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (2)
Urinary frequency (Renal and urinary disorders) | 1 (1)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Laryngeal edema (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Rash acneiform (Skin and subcutaneous tissue disorders) | 1 (1)
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 1 (2)
Hypertension (Vascular disorders) | 1 (7)
Hypotension (Vascular disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-05-07): https://cdn.clinicaltrials.gov/large-docs/01/NCT02892201/Prot_SAP_000.pdf
  • Informed Consent Form (2019-10-15): https://cdn.clinicaltrials.gov/large-docs/01/NCT02892201/ICF_001.pdf